CLINICAL TRIAL: NCT04807582
Title: Determining the Magnitude of Early Steps of Fatty Acid Oxidation in Cerebral Metastases Using [18F]FPIA PET/MRI
Brief Title: Measuring Fatty Acid Oxidation in Cerebral Metastases Using [18F]FPIA
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 19CX5551
Record Dates: First submitted 2021-03-11; First posted 2021-03-19 (Actual); Results first posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Cerebral Metastases
Keywords: PET/MRI; Fatty Acid Oxidation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample taken for carnitine analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients With Radiological Evidence of IMD That Are Treatment Naive.: Participants with radiological evidence of intracranial metastatic disease (IMD) on standard of care contrast-enhanced magnetic resonance imaging (CE-MRI) that were treatment-naive at the time of enrolment/[18F]FPIA PET-mpMRI scanning.
  Participants enrolled into the study had [18F]FPIA positron emission tomography-multiparametric magnetic resonance imaging (PET-mMRI) scan(s) performed at the Invicro, Centre for Imaging Sciences. A single intravenous dose of [18F]FPIA (maximum, 370MBq) was administered to the participant followed by a whole brain dynamic PET-MRI scan over 66 minutes.
  Interventions: Other: [18F]FPIA PET/MRI
- Patients With Radiological Evidence of IMD That Had Completed Stereotactic Radiosurgery.: Participants with radiological evidence of intracranial metastatic disease (IMD) on standard of care contrast-enhanced magnetic resonance imaging (CE-MRI) that had completed stereotactic radiosurgery (SRS) (+/- combination therapy) within 4-8 weeks of [18F]FPIA PET-mMRI.
  Participants enrolled into the study had [18F]FPIA positron emission tomography-multiparametric magnetic resonance imaging (PET-mMRI) scans performed at the Invicro, Centre for Imaging Sciences. A single intravenous dose of [18F]FPIA (maximum, 370MBq) was administered to the participant followed by a whole brain dynamic PET-MRI scan over 66 minutes.
  Interventions: Other: [18F]FPIA PET/MRI

INTERVENTIONS:
Other: [18F]FPIA PET/MRI — 18F-fluoropivalate tracer injection followed by PET/MRI scan
  Other Names: Imaging Scan

SUMMARY:
Cerebral metastases represent a significant problem for oncological management. It is estimated that 20-40% of patients with cancer will develop metastatic cancer to the brain during the course of their illness. 18F-fluoropivalate ([18F]FPIA) is a new tracer that images short chain fatty acid (SCFA) uptake in tumours, a key component of fatty acid oxidation.

The aim of this study is to quantify the degree of early step fatty acid oxidation in cerebral metastases as imaged by [18F]FPIA Positron Emission Tomography (PET)/Magnetic Resonance Imaging (MRI).

The investigators hypothesise that FPIA uptake will be higher in metastases that are treatment naïve compared to those that have undergone treatment, in keeping with viable tumour cells having a high propensity to generate ATP and NADPH via fatty acid oxidation under bioenergetic stress.

DETAILED DESCRIPTION:
24 evaluable patients with radiological evidence of cerebral metastases on MRI will be enrolled into the study (12 who are treatment naïve + 12 who have completed Stereotactic Radiosurgery (SRS)+/- combination therapy). The patients invited to participate in the study will provide written informed consent. [18F]FPIA PET/MRI imaging will only be performed once patients have satisfied the inclusion and exclusion criteria. Once these have been satisfied, eligible patients will proceed to [18F]FPIA PET/MRI.

On the day of imaging the patients will undergo a blood test to measure plasma concentrations of carnitine (approximately 6mls). During the scan, a single dose of [18F]FPIA (maximum, 370 MBq) IV will be administered to the participant followed by a whole brain dynamic PET/MRI scan over 66 minutes. During the MRI sequences, the patient will receive a 2 stage IV bolus of Gadolinium contrast medium administered through a peripheral venous cannula.

ELIGIBILITY:
Inclusion Criteria:

A) Treatment naïve

or

B) SRS+/- combination treated - Patients that have completed the SRS part of a combination regime enabling a 4-8 week post-SRS treatment PET/MRI scan.

and

C) That fulfil the following criteria:

1. Age ≥18.
2. Target metastases size ≥ 1cm.
3. WHO performance status 0 - 2.
4. If female, the subject is either post-menopausal (at least 1 year), or surgically sterilized (has had a documented bilateral oophorectomy and/or documented hysterectomy for at least 2 years), or if of childbearing potential, must have a negative urine beta human chorionic gonadotropin (beta-hCG) pregnancy test done prior to tracer administration.
5. The subject is able and willing to comply with study procedures, and signed and dated informed consent is obtained.
6. The subject has a satisfactory medical history as judged by the investigator with no significant co-morbidities.
7. The subject's clinical and laboratory tests are within normal limits and/or considered clinically insignificant.

Exclusion Criteria:

1. The subject is pregnant or lactating.
2. Any other chronic illness that will or musculoskeletal condition that would not allow comfortable performance of a PET study.
3. Prior use within 14 days of enrolment or concurrent therapy with any other investigational agent.
4. Unsatisfactory renal function (eGFR<30).
5. The subject has non-MRI compatible devices (e.g.a pacemaker, an implantable cardioverter-defibrillator (ICD), a nerve stimulator, a cochlear implant or a drug pump) or implanted material (e.g. non-MRI compatible sternal wires, biostimulators, metals or alloys).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with radiological evidence of cerebral metastases on MRI that are either treatment naïve or have been treated with SRS +/- combination therapy within 4-8 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-03-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Islam S, Inglese M, Aravind P, Barwick TD, Mauri F, McLeavy L, Arstad E, Wang J, Puccio I, Hung L, Lu H, O'Neill K, Waldman AD, Williams M, Aboagye EO. A hybrid [18F]fluoropivalate PET-multiparametric MRI to detect and characterise brain tumour metastases based on a permissive environment for monocarboxylate transport. Eur J Nucl Med Mol Imaging. 2025 Jun;52(7):2290-2306. doi: 10.1007/s00259-025-07118-0. Epub 2025 Feb 7. PMID 39915301

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was open to recruitment from Intervention: Administration of [18F]FPIA followed by the performance of a positron emission tomography-multiparametric magnetic resonance imaging (PET-mMRI) performed at Invicro, Centre for Imaging Sciences, Burlington Danes, Imperial College London (Hammersmith Hospital Campus), Du Cane Road, London, W12 0NN.
  The aim of the study was to quantify the degree of early step fatty acid oxidation in cerebral metastases as imaged by [18F]FPIA PET-mMRI.
Period: Overall Study
Arm/Group | Patients With Radiological Evidence of IMD That Are Treatment Naive. | Patients With Radiological Evidence of IMD That Had Completed Stereotactic Radiosurgery.
Started | 12 | 10
Completed | 12 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Patients With Radiological Evidence of IMD That Are Treatment Naive.: Participants with radiological evidence of intracranial metastatic disease (IMD) on standard of care contrast-enhanced magnetic resonance imaging (CE-MRI) that were treatment-naive for their IMD at the time of enrolment/[18F]FPIA positron emission tomography-multiparametric magnetic resonance imaging (PET-mpMRI).
  Participants enrolled into the study had an [18F]FPIA PET-mpMRI scan performed at the Invicro, Centre for Imaging Sciences. A single intravenous dose of [18F]FPIA (maximum, 370MBq) was administered to the participant followed by a whole brain dynamic PET-MRI scan over 66 minutes.
- Patients With Radiological Evidence of IMD That Had Completed Stereotactic Radiosurgery.: Participants with radiological evidence of intracranial metastatic disease (IMD) on standard of care contrast-enhanced magnetic resonance imaging (CE-MRI) that had completed stereotactic radiosurgery (SRS) (+/- combination therapy) within 4-8 weeks of [18F]FPIA positron emission tomography multiparametric magnetic resonance imaging (PET-mpMRI).
  Participants enrolled into the study had an [18F]FPIA PET-mpMRI scans performed at the Invicro, Centre for Imaging Sciences. A single intravenous dose of [18F]FPIA (maximum, 370 MBq) was administered to the participant followed by a whole brain dynamic PET-MRI scan over 66 minutes.
- Total: Total of all reporting groups
Arm/Group | Patients With Radiological Evidence of IMD That Are Treatment Naive. | Patients With Radiological Evidence of IMD That Had Completed Stereotactic Radiosurgery. | Total
Number analyzed (Participants) | 12 | 10 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 6 | 10
  >=65 years | 8 | 4 | 12
Age, Continuous [Median (Full Range); unit: years] | 67.5 [54 to 77] | 62.5 [46 to 66] | 64 [46 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 7 | 10
  Male | 9 | 3 | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Extracranial tumour of origin [Count of Participants; unit: Participants]
  Breast | 2 | 3 | 5
  Lung | 8 | 6 | 14
  Melanoma | 1 | 1 | 2
  Colorectal | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Quantitative Measurement of [18F]FPIA Uptake Within the Cerebral Metastases of Treatment naïve Patients.
Description: Standardised uptake value (SUV) at 60 minutes post-injection of [18F]FPIA assessed using PET/MRI. SUV is a semiquantitative measurement of radiotracer uptake in tissue. It is a ratio of tissue radioactivity concentration at a point in time within a specific region of interest and the injected dose of radioactivity per kilogram of the patient's body weight. SUVmax is the highest SUV value within a region of interest.
Time Frame: On the scan day up to 60 minutes
Measure: Mean (Standard Deviation); unit: SUV_max (kBq/L/kBq/g)
Units Other Than Participants: Lesions
Groups:
- [18F]FPIA PET-mMRI Scans Performed on Patients With Treatment-naive IMD on CE-MRI.: Participants with radiological evidence of intracranial metastatic disease (IMD) on standard of care contrast-enhanced magnetic resonance imaging (CE-MRI) that were treatment-naive for their IMD at the time of enrolment/[18F]FPIA PET-mMRI scan.
  Participants enrolled into the treatment-naive cohort that went onto have stereotactic radiosurgery (SRS) could also provide written informed consent to be scanned within the 4-8 weeks post-SRS cohort.
  Participants enrolled into the study had either one or two [18F]FPIA positron emission tomography-multiparametric magnetic resonance imaging (PET-mMRI) scans performed at the Invicro, Centre for Imaging Sciences. A single intravenous dose of [18F]FPIA (maximum, 370MBq) was administered to the participant followed by a whole brain dynamic PET-MRI scan over 66 minutes.
Arm/Group | [18F]FPIA PET-mMRI Scans Performed on Patients With Treatment-naive IMD on CE-MRI.
Number analyzed (Participants) | 12
Number analyzed (Lesions) | 17
SUV_max (kBq/L/kBq/g)
  T1 mask | 1.54 (0.41)
  SUV40 mask | 1.47 (0.33)
  SUV30 mask | 1.48 (0.33)

2. Primary Outcome: Quantitative Measurement of [18F]FPIA Uptake Within the Cerebral Metastases of Patients Treated With Stereotactic Radiosurgery (SRS).
Description: as for outcome 1
Time Frame: On the scan day (4-8 weeks post-SRS treatment)
Measure: Mean (Standard Deviation); unit: SUVmax (kBq/L/kBq/g)
Units Other Than Participants: Lesions
Groups:
- [18F]FPIA PET-mMRI Scans Performed on Patients With IMD on CE-MRI That Had Undergone SRS Treatment.: Participants with radiological evidence of intracranial metastatic disease (IMD) on standard of care contrast-enhanced magnetic resonance imaging (CE-MRI) that had completed stereotactic radiosurgery (SRS) (+/- combination therapy) within 4-8 weeks of [18F]FPIA PET-mMRI.
  Participants enrolled into the study had either one or two [18F]FPIA positron emission tomography-multiparametric magnetic resonance imaging (PET-mMRI) scans performed at the Invicro, Centre for Imaging Sciences. A single intravenous dose of [18F]FPIA (maximum, 370MBq) was administered to the participant followed by a whole brain dynamic PET-MRI scan over 66 minutes.
Arm/Group | [18F]FPIA PET-mMRI Scans Performed on Patients With IMD on CE-MRI That Had Undergone SRS Treatment.
Number analyzed (Participants) | 10
Number analyzed (Lesions) | 18
SUVmax (kBq/L/kBq/g)
  T1 mask | 1.45 (0.65)
  SUV40 mask | 1.15 (0.56)
  SUV30 mask | 1.17 (0.54)

3. Secondary Outcome: Distribution of [18F]FPIA Uptake in Lesions Which Have Undergone Treatment, With Those That Are Treatment naïve.
Description: Tumour-to-contralateral white matter (CWM) ratio (TBR) 60 minutes post-injection of [18F]FPIA using PET/MRI.
  Regions of interest for quantification were identified by an experienced neuroradiologist. For each subject, two volumes of interest (VOI) were created. A VOI was drawn around the lesion, plus a contralateral VOI of the same volume in healthy brain was measured for comparison using a T1-MRI mask, SUV30 mask and SUV40 mask.
  The maximum standardised uptake value (SUVmax) of [18F]FPIA within the tissues was calculated using the last PET frame at 60 minutes. SUV30 and SUV40 masks (30 and 40% of the SUVmax value at 60 minutes) were derived to determine image overlap.
Time Frame: On the scan day (4-8 weeks post-SRS treatment)
Measure: Mean (Standard Deviation); unit: TBRmax
Units Other Than Participants: Lesions
Arm/Group | [18F]FPIA PET-mMRI Scans Performed on Patients With Treatment-naive IMD on CE-MRI. | [18F]FPIA PET-mMRI Scans Performed on Patients With IMD on CE-MRI That Had Undergone SRS Treatment.
Number analyzed (Participants) | 12 | 10
Number analyzed (Lesions) | 17 | 18
TBRmax
  T1 mask | 3.75 (1.16) | 3.97 (1.82)
  SUV40 mask | 3.71 (1.21) | 3.85 (1.99)
  SUV30 mask | 3.73 (1.19) | 3.90 (1.94)

ADVERSE EVENTS:
Time Frame: All adverse events were reported that had taken place up to 24 hours post injection of [18F]FPIA.
Groups:
- Patients With Radiological Evidence of IMD That Are Treatment Naive.: Participants with radiological evidence of intracranial metastatic disease (IMD) on standard of care contrast-enhanced magnetic resonance imaging (CE-MRI) that were treatment-naive for their IMD at the time of enrolment/[18F]FPIA positron emission tomography-multiparametic magnetic resonance imaging (PET-mpMRI) scanning.
  Participants enrolled into the study had an [18F]FPIA PET-mpMRI scan performed at the Invicro, Centre for Imaging Sciences. A single intravenous dose of [18F]FPIA (maximum, 370MBq) was administered to the participant followed by a whole brain dynamic PET-MRI scan over 66 minutes.
- Participants With Radiological Evidence of IMD That Had Completed SRS.: Patients with radiological evidence of intracranial metastatic disease (IMD) on standard of care contrast-enhanced magnetic resonance imaging (CE-MRI) that had completed stereotactic radiosurgery (SRS) (+/- combination therapy) within 4-8 weeks of [18F]FPIA positron emission tomography-multiparametric magnetic resonance imaging (PET-mpMRI).
  Participants enrolled into the study had an [18F]FPIA PET-mpMRI scan performed at the Invicro, Centre for Imaging Sciences. A single intravenous dose of [18F]FPIA (maximum, 370MBq) was administered to the participant followed by a whole brain dynamic PET-MRI scan over 66 minutes.
Arm/Group | Patients With Radiological Evidence of IMD That Are Treatment Naive. | Participants With Radiological Evidence of IMD That Had Completed SRS.
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/10
Other Adverse Events (participants affected / at risk) | 0/12 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-08): https://cdn.clinicaltrials.gov/large-docs/82/NCT04807582/Prot_SAP_000.pdf